CLINICAL TRIAL: NCT07335133
Title: Short- and Medium-term Postoperative Complications of Ankle Arthroscopy
Brief Title: Postoperative Complications of Ankle Arthroscopy
Acronym: ARTHRO2025
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Wayan HEBRARD, Principal Investigator, Clinique Saint Jean, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-A02186-43
Record Dates: First submitted 2026-01-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ankle Injuries and Disorders; Surgery Complications
MeSH Terms: conditions — Ankle Injuries; Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of patients who underwent ankle arthroscopy (Other)
  Interventions: Other: Physical therapy and surgery tests and scores

INTERVENTIONS:
Other: Physical therapy and surgery tests and scores — Additional physical therapy and surgery tests and scores are performed on patients.

SUMMARY:
The goal of this clinical trial is to describe complications that occurred in the year following surgery, based on follow-up surgical consultations and physical therapy sessions.

The target population is any adult patient who has undergone ankle surgery performed under arthroscopy.

Primary outcome is description of all complications occurring within one year following ankle arthroscopy. This description will be based on clinical and functional examinations performed by surgeons and physical therapists.

Participants will be regularly monitored by the surgeon and physical therapist (15 days postoperative, 3 months, 6 months, and 1 year).

They will complete self-assessment questionnaires and undergo functional physical therapy tests, including ALR RSI, FAAM AVQ, FAAM Sport, CAIT, and Ankle Go.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who has been informed and has signed the consent form
* Patient scheduled for arthroscopic ankle surgery.
* Patient affiliated with or covered by a health insurance plan

Exclusion Criteria:

* Recent traumatic injury (less than 1 month old), physical therapy assessment impossible
* Inability to follow up for up to one year
* Patient under legal protection
* Pregnant woman, patient under guardianship or conservatorship
* Patient who has already undergone ankle surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Complications occurring within one year following ankle arthroscopy | One year
  Description of all complications occurring within one year following ankle arthroscopy. This description will be based on clinical and functional examinations performed by surgeons and physical therapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St jean sud de france, Montpellier, France

IPD SHARING:
Plan to Share IPD: No